CLINICAL TRIAL: NCT01734122
Title: Stereotactic Radiosurgery for Essential Tremor and Parkinsonian Tremor
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Austin Kirschner, Associate Professor, Vanderbilt University Medical Center
Other Study IDs: 120632
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Tremor; Essential Tremor; Parkinson Disease; Radiosurgery; Quality of Life
Keywords: Stereotactic Radiosurgery; Essential Tremor; Parkinsonian Tremor; Quality of Life; Severity of Tremor
MeSH Terms: conditions — Tremor; Essential Tremor; Parkinson Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Essential Tremor: Patients with severe, medication-refractory Essential Tremor
  Interventions: Other: Questionnaires / Observational Assessments
- Parkinsonian Tremor: Patients with severe, medication-refractory, tremor-dominant Parkinsons
  Interventions: Other: Questionnaires / Observational Assessments

INTERVENTIONS:
Other: Questionnaires / Observational Assessments — Includes QUEST, PDQ-39, FTM, and Neuropsych evaluation

SUMMARY:
The purpose of this study is to determine the changes in quality of life and degree of tremor for patients with essential tremor or Parkinsonian tremor who are treated by stereotactic radiosurgery (SRS). This is a questionnaire-based study. Please see Detailed Description below for more information.

DETAILED DESCRIPTION:
Tremor is the most common of all movement disorders. Patients with essential tremor (ET) or Parkinsonian tremor (PT) may be severely disabled by their tremor. When the tremor is inadequately controlled by medications, surgical options are often offered. However, some patients may prefer a noninvasive treatment approach and some patients are not surgical candidates for medical reasons.

Stereotactic radiosurgery (SRS) is a treatment that uses high-energy highly-focused radiation (X-rays) to destroy a tiny region in the brain that causes tremor to occur. This region is known as the ventral intermedius nucleus of the thalamus and is the same area targeted by surgical deep brain stimulator (DBS) treatment or neurosurgical operation (thalamotomy). Multiple case series publications using Gamma Knife stereotactic radiation have been reported that show stereotactic radiosurgery is safe and effective treatment for ET and PT, making it a standard treatment for inoperable and inadequately controlled tremor patients. However, radiation treatment by linear accelerator machines are much more common than Gamma Knife treatment machines in the United States, and there are no reports of large series of ET and PT patients treated using linear accelerator-based SRS using a noninvasive mask-based targeting system.

This clinical trial asks the question of whether linear accelerator-based SRS is as safe and effective as that reported for Gamma Knife procedures, and whether it is a valid alternative to surgical thalamotomy or implantation of a deep brain stimulator (DBS) device. The primary measurements are quality of life related to tremor before and after stereotactic radiosurgery treatment, and secondary measurements are degree of tremor severity and usage of tremor-related medications.

Stereotactic Radiosurgery (SRS) is a standard-of-care treatment for patients with severe tremor. This clinical trial is a questionnaire-based trial that only involves completion of 2 questionnaires at the consultation appointments with neurology and radiation oncology. The questionnaires only take a few minutes and will provide us with valuable information about how severe the patient's tremor is before and after SRS treatment at 3-month intervals for 1 year. Currently we are only performing SRS treatment on one side of the brain (effects one side of the body) so the side with the worst tremor is treated.

Financial: All associated steps listed below are considered the Standard of Care to receive SRS treatment for tremor and are billed to the patient's insurance per the usual routine. Patients can receive this treatment without participating in the clinical trial questionnaires. There is no financial support, no compensation, and no travel stipend available to patients who participate in this trial.

What to expect:

1. All patients interested in SRS treatment for tremor must be evaluated by a movement disorder neurologist. The neurologist will assess the severity of the tremor. Your primary physician or outside neurologist must make a referral to the Vanderbilt Movement Disorder Clinic for initial assessment. For clinical trial participation, a questionnaire will be completed as a baseline measurement (this takes a few minutes). If the patient is an appropriate candidate for SRS and there may be additional evaluations and discussion with the entire Movement Disorder group at monthly meetings.

   ** Please note: for Parkinson's disease patients, please come to the neurology evaluation "functionally off medication", which means do NOT take the morning dose of Parkinson's related medications.
2. The patient will undergo a neuropsychological evaluation prior to SRS treatment, which is the standard of care for patients considering DBS or SRS treatment.
3. The patient will meet with a neurosurgeon who will be involved in the SRS planning and procedure.
4. Patients referred for SRS treatment will be evaluated by a radiation oncologist, Dr. Austin Kirschner or Dr. Anthony Cmelak. At this appointment, discussion will include descriptions of the procedure in detail and review of the risks and benefits of treatment. For clinical trial participation, a questionnaire will be completed as a baseline assessment of the patient's tremor-related quality of life (this takes a few minutes).
5. If the patient chooses to proceed with SRS, in the department of radiation oncology a tight-fitting thermal plastic mask will be custom made to fit around the patient's head and a CT scan of the head will be performed in radiation oncology. This step takes about 45 minutes.
6. A specialized MRI of the brain will be obtained for treatment planning. This step takes about 1 hour.
7. Approximately 2 weeks after completing all the consultation appointments and obtaining the imaging for treatment planning, the single stereotactic radiation treatment will be performed. The SRS procedure takes approximately 2.5 hours. It is entirely outpatient and does not require anesthesia. The procedure is noninvasive and painless (X-ray treatment). During the entire treatment, the head is held tightly in the plastic mask. Oral anti-anxiety medication may be given to relax the patient.

   Follow-up:
8. At 3 month intervals for 1 year, the patient will have follow-up appointments with radiation oncology and neurology. A brain MRI may be performed at some of these intervals to document the treatment effect on the brain tissue. For participation in the clinical trial, at these follow-up appointments the quality of life questionnaire will be completed at the radiation oncology visit and the severity of tremor questionnaire will be completed at the neurology visit .
9. At 6 months after SRS treatment, a neuropsychological evaluation will be performed.

All patients interested in stereotactic radiosurgery (SRS) or participating in this questionnaire-based clinical trial should feel free to call the contact phone numbers listed below or have their physician refer the patient for consultation with the Movement Disorder Clinic in the neurology department at Vanderbilt.

ELIGIBILITY:
Inclusion Criteria:

* Must be certified by a neurologist as having essential tremor or Parkinsonian tremor that is insufficiently controlled by medication alone.
* Preference to receive radiation treatment for tremor treatment, rather than surgical DBS implantation or surgical thalamotomy
* At least 18 years old

Exclusion Criteria:

* Contraindications to cranial radiation (such as prior radiation to the thalamus)
* Inability to have a MRI of the brain
* Prior surgical thalamotomy treatment (but contralateral deep brain stimulator [DBS] is permitted)
* Estimated life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This trial enrolls persons with essential tremor or Parkinsonian tremor that is inadequately controlled by medications.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-02-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Tremor-related Quality of Life | 1 year
  The tremor-related quality of life for each patient will be assessed by self-assessment questionnaire at 3 month intervals for 1 year after treatment by stereotactic radiation.

SECONDARY OUTCOMES:
Severity of Tremor | 1 year
  The severity of tremor will be assessed by objective measure (Fahn-Tolosa-Marin tremor rating scale) at 3 month intervals for 1 year following the stereotactic radiation treatment.
Neuropsychological Assessment | Baseline and 6 months post-treatment
  All patients will undergo a neuropsychological assessment (1-2 hr examination) at baseline and at 6 months post-treatment. This will assess any unanticipated changes in neuropsychological brain function.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luo G, Neimat JS, Cmelak A, Kirschner AN, Attia A, Morales-Paliza M, Ding GX. Margin of error for a frameless image guided radiosurgery system: Direct confirmation based on posttreatment MRI scans. Pract Radiat Oncol. 2017 May-Jun;7(3):e223-e231. doi: 10.1016/j.prro.2016.08.006. Epub 2016 Aug 20. PMID 27720703
- [Background] Khattab MH, Cmelak AJ, Sherry AD, Luo G, Wang L, Yu H, Hedera P, Phibbs FT, Lindsell CJ, Neimat J, Kirschner AN. Noninvasive Thalamotomy for Refractory Tremor by Frameless Radiosurgery. Int J Radiat Oncol Biol Phys. 2022 Jan 1;112(1):121-130. doi: 10.1016/j.ijrobp.2021.08.021. Epub 2021 Aug 25. PMID 34454047
- [Background] Luo G, Cameron BD, Wang L, Yu H, Neimat JS, Hedera P, Phibbs F, Bradley EB, Cmelak AJ, Kirschner AN. Targeting for stereotactic radiosurgical thalamotomy based on tremor treatment response. J Neurosurg. 2021 Oct 29;136(5):1387-1394. doi: 10.3171/2021.7.JNS21160. Print 2022 May 1. PMID 34715657
- See also: Find a Clinical Trial — http://www.vicc.org/ct/